CLINICAL TRIAL: NCT01699321
Title: Promoting Physical Activity in Black Barbershops
Brief Title: FITShop: Promoting Physical Activity in Black Barbershops
Acronym: FITShop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Central University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-1903; 1U54CA156733 (NIH)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Physical Activity
Keywords: physical activity; barbershop; cancer prevention; exercise; men's health; African American men
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Your Move (physical activity) (Experimental): The Your Move intervention is a multi-level, theory and evidence-based intervention that will include the following components: monthly handbills with community resources, newsletters, contests (shop and customer level), tailored health feedback report, and monthly phone calls from the research team.
  Interventions: Behavioral: Your Move (physical activity)
- Your Money (financial empowerment) (Other): The Your Money program is an attention control intervention. Owners and barbers will receive 3 workshops that focus on financial health. Customers will receive monthly handbills and newsletters about different financial health topics.
  Interventions: Other: Your Money (financial empowerment)

INTERVENTIONS:
Behavioral: Your Move (physical activity) — Materials that are provided will aim to increase a participant's minutes of physical activity.
  Arms: Your Move (physical activity)
Other: Your Money (financial empowerment) — Materials that are provided to participants will direct them to resources for financial health.
  Arms: Your Money (financial empowerment)

SUMMARY:
Physical activity has been proven to reduce the risk of cancer. The North Carolina FITShop research study will test the effectiveness of a program aimed at increasing physical activity among African American men. Approximately 14 barbershops and 560 shop customers within Orange, Durham, Chatham, Alamance, and Wake counties will be enrolled into this research study. If FITShop is effective, we will share our results throughout North Carolina and nationally.

DETAILED DESCRIPTION:
Black men suffer disproportionately higher rates of nearly all disease categories, including cancer --the leading cause of death in North Carolina. An estimated 50% of cancer is preventable with lifestyle modifications such as increasing physical activity (PA), eliminating tobacco use/exposure and maintaining a healthy weight. Evidence suggests that physical activity can reduce risk to several types of cancer. Innovative ways to reach Black men with effective health promotion interventions are needed. Barbershops represent one place where Black men can be reached, but have not been utilized as settings for intervening to promote physical activity. An experienced, interdisciplinary, partnership between community members (barbershop owners, barbers and their customers) and researchers from UNC Chapel Hill/Lineberger Comprehensive Cancer Center and the Gillings School of Global Public Health, and North Carolina Central University are conducting a two-phase outreach study to bridge this gap. Phase 1 is a series of inter-related formative research studies (in-depth interviews with barbers/owners; observations in shops; focus groups with customers) leading to the development of a theory and evidence-guided, multi-level physical activity intervention (FITShop) designed to increase PA among Black men in barbershops. Using Phase 1 results, Phase 2 is a two-arm, group randomized, initial efficacy trial of the FITShop intervention in 14 Black barbershops with 40 customers per shop (n=560 total). Customers in Arm 1 (7 shops, 280 customers) will receive the FITShop intervention which includes barber training, PA contest in the shop, use of pedometers, community connections and personal feedback plus recommendations for PA. Customers in Arm 2 (7 shops, 280 customers) will receive a Financial Empowerment (FE) attention-control intervention that mimics exposure amount without influencing the primary outcome. Consistent with community-based participatory research principles, an Advisory Board will guide all aspects of the study planning, development, implementation and analysis of results. The primary outcome (physical activity) will be measured via accelerometer using a 7-day protocol and with self-report questionnaires at baseline and 6 months using a previously tested protocol with Black men recruited from barbershops. All primary/secondary outcomes will be measured on all customers at an assessment event/via questionnaire prior to randomization (and at 6 mo) using standardized, previously tested protocols. Process evaluation will assess dose of intervention delivered, received, fidelity, as well as reach, adoption and representativeness at the customer, barber and barbershop levels. Since barbershops are located in all communities, if effective, this intervention has promise for dissemination & sustainability.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* African American
* Male
* Regular customer of the barbershop

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in physical activity measures | Baseline and 6 months
  Minutes of physical activity will be self-reported along with physical activity status, self-efficacy, barriers, etc. Accelerometers will be given at baseline and the 6 month follow-up.

SECONDARY OUTCOMES:
Change in smoking status | Baseline and 6 months
  Self-reported smoking status (y/n)
Change in weight/BMI | Baseline and 6 months
  Participants weight will be measured at baseline and 6 months. Their BMI will be calculated
Change in waist circumference | Baseline and 6 months
  Participant's waist circumference will be measured at baseline and 6 months.
Change in resting heart rate | Baseline and 6 months
  Participant's resting heart rate will be measured at baseline and 6 months.
Change in blood pressure | Baseline and 6 months
  Participant's blood pressure will be measured at baseline and 6 months.
Change in aerobic fitness level | Baseline and 6 months
  Participant's aerobic fitness level will be measured using a step test at baseline and 6 months.
Change in psycho-social variables | Baseline and 6 months
  Participant's will self-report psycho-social variables at baseline and 6 months.
Change in barber-customer interactions | Baseline and 6 months
  Research team will conduct shop observations at baseline and 6 months.
Change in barbershop characteristics | Baseline and 6 months
  Barbershop characteristics will be reported through environmental scans of the shop and informational interviews with the owners and barbers.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Linnan, ScD, CHES, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - North Carolina Central University, Durham, North Carolina